CLINICAL TRIAL: NCT06524531
Title: Safety and Efficacy of Pulsed RF Neuromodulation and Leukocyte-Rich PRP for the Treatment of Refractory Low Back Pain Due to Multifidus Dysfunction
Brief Title: Pulsed RF Neuromodulation and Leukocyte-Rich PRP for Refractory Low Back Pain
Acronym: Multifidus
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Iffat Anwar Medical Complex (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IAMC003
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Multi-Organ Disorder
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Pulsed RF Neuromodulation: Administered to the L2 and L3 segments bilaterally for 6 minutes each.
  Leukocyte-Rich PRP Injection: Injected into the multifidus muscle. Physiotherapy: Standard physiotherapy regimen.
  Interventions: Procedure: Pulsed RF Neuromodulation; Biological: Leukocyte-Rich PRP Injection
- Control Group (Experimental): Physiotherapy: Standard physiotherapy regimen only
  Interventions: Procedure: Physiotherapy Alone

INTERVENTIONS:
Procedure: Pulsed RF Neuromodulation — RF neuromodulation will be applied to the L2 and L3 segments bilaterally. Each segment will receive treatment for 6 minutes, either sequentially or simultaneously on both sides.
  Arms: Experimental Group
Biological: Leukocyte-Rich PRP Injection — Leukocyte-rich PRP will be prepared from the patient's blood and injected into the multifidus muscle at the L2 and L3 levels.
  Arms: Experimental Group
Procedure: Physiotherapy Alone — Standard physiotherapy regimen tailored to each participant's needs. This may include exercises to improve flexibility, strength, and endurance of the back muscles, as well as education on posture and body mechanics.
  Arms: Control Group

SUMMARY:
This clinical trial aims to check the safety and efficacy profile of pulsed radiofrequency (RF) neuromodulation combined with leukocyte-rich platelet-rich plasma (PRP) injections for the treatment of refractory low back pain due to multifidus dysfunction. The trial will compare two groups: one receiving standard physical therapy and the other receiving pulsed RF neuromodulation and physiotherapy.

DETAILED DESCRIPTION:
Low back pain is a common condition, often associated with multifidus muscle dysfunction, which can result from aging, obesity, or limited movement. This dysfunction is characterized by fatty infiltration and loss of muscle function. Surgical procedures involving posterior or transpedicular screw insertion can exacerbate this issue by damaging the multifidus muscle, leading to persistent pain.

This study will investigate the effects of pulsed RF neuromodulation on the L2 and L3 segments bilaterally, with each side receiving treatment for 6 minutes. In addition, leukocyte-rich PRP will be injected into the multifidus muscle, and patients will undergo a physiotherapy regimen. The primary outcomes will be compared with those of a control group receiving only physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Refractory low back pain due to multifidus dysfunction.
* Pain persisting for more than 6 months despite conventional treatments.
* Ability to provide informed consent.

Exclusion Criteria:

* Previous spinal surgery within the last year.
* Current use of systemic steroids or immunosuppressive medications.
* Known bleeding disorders or anticoagulant therapy.
* Pregnancy or lactation.
* Severe psychiatric or cognitive disorders.
* Any Congenital or Non-congenital disorders

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-07-10 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain Visual Analog Scale (0-10) | 2 Weeks
  Change in pain intensity from baseline
Pain Visual Analog Scale (0-10) | 3 Months
  Change in pain intensity from baseline
Pain Visual Analog Scale (0-10) | 6 Months
  Change in pain intensity from baseline
Pain Visual Analog Scale (0-10) | 1 Year
  Change in pain intensity from baseline
Oswestry Disability Index (0-50) | 2 Weeks
  Change in disability index from baseline
Oswestry Disability Index (0-50) | 3 Months
  Change in disability index from baseline
Oswestry Disability Index (0-50) | 6 Months
  Change in disability index from baseline
Oswestry Disability Index (0-50) | 1 Year
  Change in disability index from baseline
Hospital Anxiety and Depression Scale (0-14) | 2 Weeks
  Change in anxiety and depression levels from baseline
Hospital Anxiety and Depression Scale (0-14) | 3 Months
  Change in anxiety and depression levels from baseline
Hospital Anxiety and Depression Scale (0-14) | 6 Months
  Change in anxiety and depression levels from baseline
Hospital Anxiety and Depression Scale (0-14) | 1 Year
  Change in anxiety and depression levels from baseline
Quality of Life (0-100) | 2 Weeks
  Change in Quality of life from baseline
Quality of Life (0-100) | 3 Months
  Change in Quality of life from baseline
Quality of Life (0-100) | 6 Months
  Change in Quality of life from baseline
Quality of Life (0-100) | 1 Year
  Change in Quality of life from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Iffat Anwar Medical Complex, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No